CLINICAL TRIAL: NCT00003416
Title: S9805, Phase II Study of Tandem High Dose Melphalan Supported by Peripheral Blood Stem Cell Support in Waldenstrom's Macroglobulinemia (WM)
Brief Title: S9805, High-Dose Melphalan Plus Peripheral Stem Cell Transplantation Followed by Interferon Alfa in Treating Patients With Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S9805; S9805 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-08-03 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Lymphoma
Keywords: Waldenström macroglobulinemia
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia | interventions — Filgrastim; Interferon-alpha; Dexamethasone; Melphalan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): Ind:
  dexamethasone 40 mg/d PO D1-4,9-12,17-20 q35 days x 3 cycles
  SC Collection:
  cyclophosphamide 1.5gm/m2 IV q3 hrs x 2 mesna 3 gm/m2 conIV start with cyclo GCSF 5mcg/kg/d SQ start 1 day after cyclo until WBC > 50,000/mcg
  Trans (x2):
  melphalan 100 mg/m2/d IV D-1,-2 PBSC infusion D0
  Maint:
  interferon 3 million units/m2 SQ 3x/wk
  Interventions: Biological: filgrastim; Biological: recombinant interferon alfa; Drug: dexamethasone; Drug: melphalan; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: recombinant interferon alfa
Drug: dexamethasone
Drug: melphalan
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy and kill more tumor cells. Interferon alfa may interfere with the growth of the cancer cells.

PURPOSE: Phase II trial to study the effectiveness of high-dose melphalan plus peripheral stem cell transplantation followed by interferon alfa in treating patients with Waldenstrom's macroglobulinemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess remission rates and overall and progression-free survival in patients with Waldenstrom's macroglobulinemia treated with tandem high dose melphalan supported by peripheral blood stem cell support. II. Assess the associated hematologic and nonhematologic toxicities of this regimen in these patients.

OUTLINE: Regimen A (dexamethasone induction): All patients receive high dose dexamethasone orally on days 1-4, 9-12, and 17-20; courses repeat every 35 days for a total of 3 courses. Regimen B (stem cell mobilization and collection): Following a 4-6 week break after dexamethasone induction and regardless of response or progression, patients have stem cells collected following administration of filgrastim (G-CSF) by injection; G-CSF continues until completion of stem cell collection (maximum of 6 aphereses). Regimen C (first peripheral blood stem cell transplant (PBSCT)): Regardless of disease progression, patients recovered from toxicities from dexamethasone induction and stem cell mobilization and collection, and who have adequate number of CD34 cells collected for at least 1 transplant, receive 1 dose of melphalan daily for 2 days followed by peripheral stem cell reinfusion. G-CSF is given by injection beginning on the day after peripheral stem cell reinfusion and continues until the absolute granulocyte count is greater than 1,000/mm3 on 3 consecutive days. Regimen D (second PBSCT): Patients who had adequate stem cell collection for 2 transplants during regimen B, have no evidence of disease progression after the first transplant, and have recovered from effects of previous treatment undergo a second treatment with high dose melphalan with PBSCT and G-CSF support, given 3-12 months following the first transplant. Patients who had enough cells collected for only one transplant go directly to regimen E. Regimen E (maintenance interferon alfa): Beginning 5-12 weeks after transplant and upon hematologic recovery of blood counts and other toxicities, patients with at least a partial response after high dose melphalan and PBSCT receive subcutaneous interferon alfa injections 3 times a week for 5 years or until disease progression, relapse, or toxicity. Patients are followed every month for 6 months, then every 3 months for 5 years, then annually thereafter.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study over 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Immunologically diagnosed Waldenstrom's macroglobulinemia (WM) Evaluable quantifiable IgM One of the following criteria must be met: 1) Patient demonstrates clinical symptoms such as fatigue, dizziness, visual inacuity, or hemorrhagic manifestations of WM with anemia, hyperviscosity, thrombocytopenia, or coagulopathies 2) Advanced tumor mass present involving ONE of the following: Extensive lymphadenopathy (greater than 2 cm) Hepato or splenomegaly palpable on clinical examination Marked bone marrow infiltration greater than 50% 3) Progressive disease; i.e., increase in IgM concentration by at least 50%, and/or a drop of greater than 2 g/dL in hemoglobin (in the absence of gastrointestinal bleeding), and/or a greater than 50,000/mm3 decrease in platelets

PATIENT CHARACTERISTICS: Age: Under 70 Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Not specified Renal: Not specified Cardiovascular: At least 6 months since myocardial infarction No congestive heart failure No arrhythmia refractory to therapy Ejection fraction within normal range by MUGA or ECHO Pulmonary: FEV1 at least 50% of predicted DLCO at least 50% of predicted Other: Not pregnant or nursing Effective contraception required of fertile patients No significant comorbid condition No uncontrolled life-threatening infection No uncontrolled diabetes No other malignancy within past 5 years except adequately treated basal or squamous cell skin cancer, carcinoma in situ of the cervix or adequately treated stage I or II cancer currently in remission HIV negative Hepatitis B surface antigen negative

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since chemotherapy and recovered Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since radiotherapy and recovered Surgery: Not specified

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 1998-09; Primary Completion 2000-08 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
confirmed remission rate | until death
overall survival (OS) | until death
progression free survival (PFS) | until death
toxicity | until death

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Dhodapkar, MD, Study Chair — Rockefeller University
Locations (84):
- United States (84):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Beckman Research Institute, City of Hope, Duarte, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Hospital - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington